CLINICAL TRIAL: NCT04328753
Title: The Effect of Super Oxidized Water Mouthwash on the Level of IL_1β in Gingival Crevicular Fluid and Some Clinical Periodontal Parameters for Patients With Gingivitis: Randomized Clinical Trial
Brief Title: The Effect of SOW Mouthwash on the Level of IL_1β in GCF and Some Clinical Periodontal Parameters for Patients With Gingivitis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Ali Jawad, Specialist dentist, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Baghdad University
Record Dates: First submitted 2020-03-24; First posted 2020-03-31 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Generalized Gingivitis

STUDY DESIGN:
Intervention Model Description: Forty-five adult male patients with generalized gingivitis participated in the double blinded randomized controlled parallel study divided into three groups, two mouth rinses and distilled water( negative control) used during seven days periods as adjunctive to regular mechanical oral hygiene, one group received super oxidized water mouth rinses(microsafe®) three times daily and the second group received Alcohol-free chlorhexidine 0.12% solution(kin gingival®) twice dialy and the third group received distilled water (negative control).
Who Masked: Outcomes Assessor
Masking Description: third professional person give the one of opaque coded bottle to the participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- super oxidized water group (Experimental)
  Interventions: Drug: Super Oxide water
- chlorhexidene group (Active Comparator)
  Interventions: Drug: Chlorhexidine mouthwash
- distilled water (Placebo Comparator)
  Interventions: Other: Distilled water

INTERVENTIONS:
Drug: Super Oxide water — Microsafe®, a recently available super-oxidized solution for gingival care, offers a completely improved approach for treatment of gingivitis. The neutral pH, super oxidized water was certified as an antiseptic .
  Other Names: SOW
  Arms: super oxidized water group
Drug: Chlorhexidine mouthwash — CHX is a regular bisbiguanide artificial antiseptic containing of two biguanide groups and four chlorophenyl rings linked by a hexamethylene bridge. The dicationic nature of CHX makes it interacting strongly with anions, which is related to its safety, efficacy, and side effects. It is available in three forms, digluconate, acetate and hydrochloride salts. CHX has broad spectrum antimicrobial activity
  Other Names: CHX
  Arms: chlorhexidene group
Other: Distilled water — act as a negative control in this study
  Other Names: D.W
  Arms: distilled water

SUMMARY:
Forty-five adult male patients with generalized gingivitis participated in the double blinded randomized controlled parallel study divided into three groups, two mouth rinses and distilled water( negative control) used during seven days periods as adjunctive to regular mechanical oral hygiene, one group received super oxidized water mouth rinses(microsafe®) three times daily and the second group received Alcohol-free chlorhexidine 0.12% solution(kin gingival®) twice dialy and the third group received distilled water (negative control).

The first visit included PLI measurement after that we removed the supra gingival plaque by cotton roll to avoid contamination with the periopaper strip during GCF collection, then GCF collected from targeted sites(upper incisors, labial side) after that the other clinical periodontal parameters ( GI and BOP) were measured and then scaling was done after sample collection because of gingival bleeding which occur during scaling then inform the patient to use the coded bottle which gave to the participant by the assistant not involve in the study so the researcher did not know the type of mouthwash that was given to the participant( CHX twice daily while SOW three times daily) .The mouthwashes was given for one week with routine mechanical dental home care(brushing and flossing).The codded bottle was gave randomly by a decision on that day for example on Sunday we gave all the participants code 1 and on other days we gave to other participants code 2 or code 3.

In the second visit the PLI was measured first , then the sample was collected from the same teeth after that the other periodontal parameters were collected again ( GI and BOP).

DETAILED DESCRIPTION:
One of the most predominant periodontal diseases is the plaque induced gingivitis. : For the past 20 years, super-oxidized solutions have been shown to be powerful antimicrobials and disinfectants via oxidative damage. The taste is better than chlorhexidine and doesn't stain the teeth. Some individuals experience a slight burning sense in the mouth when gargling. They should be taught to spit out the solution. The burning sensation then dispels. Microsafe®, a recently presented super-oxidized solution for gingival care, offers a completely improved approach to treatment of gingivitis. The neutral pH, super oxidized water was certified as an antiseptic in México in 2004. Animal tests were initially conducted to show that Microsafe® does not make irritation or sensitization in skin and mucosa. Interleukin 1 beta is one from interleukin family and it is released by many cells such as macrophage to control immune response.

Aims of the study

The aim of the study is to determine the effect of super oxidized water mouthwash on the pro inflammatory cytokines (IL_1β) in the gingival crevicular fluid and its effect on some clinical periodontal parameters (plaque index, gingival index and bleeding on probing index) compared to chlorhexidine in participants who continue to perform regular mechanical oral hygiene.

Objective To evaluate the efficacy of SOW on IL_1β by using ELISA technique Null hypothesis SOW has anti inflammatory effect by reducing IL_1β and some clinical periodontal parameters (plaque index, gingival index and bleeding on probing index) when used by the patients with regular mechanical oral hygiene.

Alternative hypothesis The effect of SOW mouth rinse(microsafe®) is less than Alcohol-free CHX 0.12% mouth rinse(kin gingival®) on the the inflammatory marker IL_1βand some clinical parameters (PI,GI and BOP).

Materials and methods

Forty-five adult male patients with generalized gingivitis participated in the double blinded randomized controlled parallel study divided into three groups, two mouth rinses and distilled water( negative control) used during seven days periods as adjunctive to regular mechanical oral hygiene, one group received super oxidized water mouth rinses(microsafe®) three times daily and the second group received Alcohol-free chlorhexidine 0.12% solution(kin gingival®) twice dialy and the third group received distilled water (negative control).

The first visit included PLI measurement after that we removed the supra gingival plaque by cotton roll to avoid contamination with the periopaper strip during GCF collection, then GCF collected from targeted sites(upper incisors, labial side) after that the other clinical periodontal parameters ( GI and BOP) were measured and then scaling was done after sample collection because of gingival bleeding which occur during scaling then inform the patient to use the coded bottle which gave to the participant by the assistant not involve in the study so the researcher did not know the type of mouthwash that was given to the participant( CHX twice daily while SOW three times daily) .The mouthwashes was given for one week with routine mechanical dental home care(brushing and flossing).The codded bottle was gave randomly by a decision on that day for example on Sunday we gave all the participants code 1 and on other days we gave to other participants code 2 or code 3.

In the second visit the PLI was measured first , then the sample was collected from the same teeth after that the other periodontal parameters were collected again ( GI and BOP).

ELIGIBILITY:
Inclusion Criteria:

* 1. patient with generalized gingivitis. 2. no antibiotic treatment during a 3-month period prior to the start of the trial.

  3. no regular medication with anti-inflammatory compounds. 4. no history of allergy to oral care products. 5. no regular use of oral antiseptics.

Exclusion Criteria:

* 1. Patients who refuse to write an informed consent form. 2. Smokers. 3. Female patients

Ages: 15 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Forty-five adult male patients with generalized gingivitis
Enrollment: 45 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-05-20 (Estimated); Study Completion 2020-06-24 (Estimated)

PRIMARY OUTCOMES:
measuring interleukin -1 beta | one week
  measure interleukin -1 beta in gingival crevicular fluid by using ELISA

SECONDARY OUTCOMES:
measuring plaque accumulation | one week
  measure plaque accumulation on the teeth by measuring the plaque index using periodontal probe
measuring gingival inflammation | one week
  measure gingival inflammation by measuring the gingival index using periodontal probe
measure the gingival sulcus erosion | one week
  measure the gingival sulcus erosion and destruction by measuring the bleeding on probing index using periodontal probe

CONTACTS AND LOCATIONS:
Locations (1):
- Baghdad university college of dentistry, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No